CLINICAL TRIAL: NCT06150313
Title: Efficacy of the Mediational Intervention for Sensitizing Caregivers - Teachers' Version (MISC-T) and Self-Administered Version (MISC-SA) to Improve the Quality of Caregivers' Interactions and Children Mental Health (MISC-SA/T Project)
Brief Title: Efficacy of the Mediational Intervention for Sensitizing Caregivers for Teachers and Self-Administered Versions
Acronym: MISC-SA/T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Autonoma de Barcelona (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Sergi Ballespí, Ph.D., Principal Investigator, Universitat Autonoma de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PID2021-125444OB-100
Record Dates: First submitted 2023-09-26; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel group, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediational Intervention for Sensitizing Caregivers, Teachers' version (MISC-T) (Experimental): MISC-T is an adaptation of MISC for trainers. The trainer is the figure who trains a caregiver to enable him/her to interact with higher quality (i.e., with more MISC components). MISC for trainers is commonly administered to groups of 6-20 trainees, either face to face or using videoconference, and consists of 8 hours of theory about MISC principles and 12 hours of practice using video feedback. Video feedback is the core component of MISC training, which aims to transfer more competency than knowledge, using ecological practice. This means using video recordings of daily interactions with a significant child and watching them together (supervisor and trainee) to enable the trainee to realize the consequences of MISC components. MISC for trainers was adapted to be administered to groups of 6-12 teachers using 4 x 2-hours theoretical sessions (8h) and 11 x 1.5-hours of practice using video-feedback.
  Interventions: Behavioral: Mediational Intervention for Sensitizing Caregivers, Teachers' version (MISC-T)
- Mediational Intervention for Sensitizing Caregivers, Self-Administered version (MISC-SA) (Experimental): This MISC version (MISC-SA) aims to transference the MISC training to wider communities by diminishing the cost of the teaching and learning. By implementing the MISC lessons in an online platform, thus allowing self-learning, the new Self-Administered version of MISC allows to obtain MISC training in 25 weekly sessions distributed across 7 months (approximately, a scholar course). In contrast to MISC-T, this version allows the simultaneous self-training of a high number of participants with very low intervention of a supervisor, which diminishes the cost. As MISC-T, MISC-SA keeps the core component of MISC trainings (video-feedback) by fostering participants to record interactions and then visualize them using guided reflection.
  Interventions: Behavioral: Mediational Intervention for Sensitizing Caregivers, Self-Administered version (MISC-SA)
- Mediational Intervention for Sensitizing Caregivers - Readings version (MISC-R) (Active Comparator): Teachers usually do not get training to improve the quality of the interactions. However, to avoid using a Waiting-List or a Placebo control group, a last version of MISC training was designed but, this time, without the core MISC component: video-feedback. MISC-Readings provides the theoretical knowledge of MISC but lacks practice and reflection of MISC components by watching once own video recorded interactions with a significant child. MISC-Readings substitutes all the practice time of the other versions (video-feedback) by readings, that is, theoretical knowledge. This assimilates this version to the 'intellectual' or more theoretical format of teachers' common training, even when it is referred to social-emotional learning.
  Interventions: Other: Mediational Intervention for Sensitizing Caregivers - Readings version (MISC-R): Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Mediational Intervention for Sensitizing Caregivers, Teachers' version (MISC-T) — This is a 36-hour group training involving 4 theoretical + 11 practice online sessions using video-feedback, the core component of MISC original trainings.
  Session 1: MISC presentation; Session 2: Bases of the interaction and MISC culture-context components; Session 3: The emotions in the interaction and MISC emotional components; Session 4: MISC cognitive components and implications for learning; Session 5: Practice with you-tube examples of interaction; Session 6: Practice with trainer's examples of video-feedback. Sessions 7 to 14: Practice with participants' video-recordings. Session 15: End of the intervention, last video-feedback training and preparing for post-assessment.
  Other Names: MISC for Trainers adapted for groups of Teachers; MISC-T
  Arms: Mediational Intervention for Sensitizing Caregivers, Teachers' version (MISC-T)
Behavioral: Mediational Intervention for Sensitizing Caregivers, Self-Administered version (MISC-SA) — This is a 36-hour individual training involving 25-weekly online, individual, self-administered 50' sessions (21h) + 4 online 1.5-hour group meetings with a supervisor (6h) and 9h of between sessions work (readings, video-recordings for later video-feedback, reflection exercises). Session 1 (Supervisor): Presentation of the MISC program; Sessions 2 to 8 (Self-Administered or SA): Theoretical bases of the MISC: Session 9 (Supervisor): Summary, online group exercises and keys for forward recordings; Sessions 10-11 (Christmas Homework): Recording daily life interactions; Sessions 12-17 (SA): guided reflection with video-feedback; Session 18 (Supervisor): Control session for doubts and video-feedback group training. Sessions 19-28 (SA): guided reflection with video-feedback. Session 29 (Supervisor): Final online video-feedback group training.
  Other Names: MISC-SA
  Arms: Mediational Intervention for Sensitizing Caregivers, Self-Administered version (MISC-SA)
Other: Mediational Intervention for Sensitizing Caregivers - Readings version (MISC-R): Treatment as Usual (TAU) — This is an equivalent 36-hour online self-administered training involving 27 x 45' individual online sessions (20.25h), mostly based on reflection exercises around brief readings, animated shorts, or pills, but not video-feedback. This is complemented with 2 x 1.5h online group face-to-face sessions with a supervisor (3h) and 13h of between-sessions work based on looking for new information, adult-child activities (but not for video-feedback) or out-of-line guided reflective exercises. Session 1 (Supervisor): group meeting for program presentation; Sessions 2-28 (Self-Administered): Online self-administered sessions doing readings or watching pills; Session 29 (Supervisor): Final doubts session to close de course.
  Other Names: MISC-R; TAU
  Arms: Mediational Intervention for Sensitizing Caregivers - Readings version (MISC-R)

SUMMARY:
OBJECTIVES: The goal of this parallel randomized controlled trial is to test the efficacy of 2 new modalities of the Mediational Intervention for Sensitizing Caregivers (MISC) in caregivers from general population, specifically, in teachers at primary school children who are also parents.

The main QUESTIONS it aims to answer are:

* Are the new versions of MISC (MISC-T for Teachers, and MISC-SA or Self-Administered) efficient to a) improve the quality of caregivers-child interaction, and b) benefit children mental health, compared with a control group defined as Treatment as Usual (TAU)?
* Is there any effect-transference to the school-setting despite the MISC is trained out of the school setting? re the new versions of the MISC efficient to benefit teachers' well-being at work in terms of lower burn-out, higher perceived self-efficacy or better classroom climate?

PARTICIPANTS will randomly receive one of the 3 versions of MISC: MISC-T (administered by videoconference in teams of 6-10 teachers), MISC-SA (self-administered by the participants in weekly sessions with Genially), and MISC-R (self-administered by the participants but mainly based in readings and cognitive exercises instead of video-feedback, the core element of MISC-T and MISC-SA).

COMPARISONS: Researchers will compare all 3 groups among them to see to what extent:

* MISC-T shows efficacy compared with MISC-R (TAU; control group)
* MISC-SA shows efficacy compared with MISC-R (TAU; control group)
* MISC-T is more efficient than MISC-SA

DETAILED DESCRIPTION:
CONTEXT: Mental health interventions are mostly provided once mental health is lost, that is, in context of psychopathology (clinical impairment). James Heckman's Equation suggests that investing in mental health before it is severely impaired would lead to high returns. We want to test: 1) to what extent is possible to transfer active ingredients for mental health from the clinical context to the community, and 2) to what extent an intervention aimed to enrich parents and teachers social-emotional skills (two of the main figures in child rearing) improves children mental health. Because this intervention aims to reach a wide community in non-clinical settings, it should be extensive (to ensure solid changes in the child environment) and cost-efficient, that is: cheaper than those individually transmitted in the classic therapist-client relationship.

METHODOLOGY: 17-month multisite, Randomized, Controlled Trial (RCT).

MEASURES OPERATIONALIZATION: It is expected that this translational intervention which aims to move factors for salutogenesis from the clinical setting to non-clinical points of the mental ill-health continuum could benefit both the caregivers who receive the intervention (who are parents and teachers as well) and the children who daily exposed to them (their own children and their school students). Caregivers' benefits are expected in terms of improved mentalizing capacities, lower stress, higher well-being and higher sense of self-efficacy both at home (parenting) and at work (school). Child's mental health is operationalized s multidimensional using: the number of symptoms, the level of role- and social functioning, and well-being. Child's benefits in terms of mentalization and pro-social behavior are also expected because of the long-term exposition to adults enriched with new social-emotional skills thanks to the intervention.

STATISTICAL ANALYSES: The analysis under the Intention-To-Treat (ITT) approach will encompass all participants subjected to random allocation, with the utilization of multiple imputation techniques to address any missing data. Estimation of parameters, accounting for the specific statistical assumptions of each model and the data's characteristics, will be carried out through the implementation of Linear Mixed-Effect Models and Structural Equation Modeling (SEM). Various R packages will be employed to execute these models, primarily "lme4" and "nlme" for linear mixed-effect models, and "lavaan" for SEM models. Concerning statistical power, a sample size of 150 participants (50 per arm) has been proposed, which exceeds the minimum of 54 participants (18 per arm) required to detect a medium effect size (Cohen's d=0.25) in the design comprising 3 arms, 3 repeated measures (pre, post, and 1 follow-up), and a power level of .95. An empirical power close to 1.00 is anticipated. Effect size measures, including Cohen's d and squared Omega statistics, will be employed.

ELIGIBILITY:
Inclusion criteria:

Teachers of school- or preschool-age children, currently teaching, who are parents (either of a school-age child (6-12 years old) or an adolescent (12-18)), or who can record interactions with a similar age close child (e.g., nephew). The "parent" condition is important because a) it allows participants to do this training with a very close child (son/daughter) with who it is easy to record daily-life interactions to then train using video-feedback, a key element in MISC (Mediational Intervention for Sensitizing Caregivers); b) because it allows a uniform measurement of the impact of parental MISC intervention in the mental health of the children currently (daily) exposed to those parents (their sons/daughters). The "teacher" condition allows to examine to what extent MISC training effects might be transferred beyond the own child (with whom the training is done: son / daughter) and can be extended to other contexts like the school setting.

1. Teachers at school- (6-12) or preschool (3-6) in active
2. Parents who have a son or daughter 6-18 years old
3. Possibilities to receive at least 1 of the 3 interventions
4. Understanding Catalan
5. Written informed content

Exclusion criteria:

1. Teachers who are not currently teaching in school or preschool degrees
2. Impossibility to record interaction with a significant child
3. Inability to attend the intervention randomly assigned

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
OMI (Observing Mediational Interaction) | Through study completion, an average of 17 months
  This is the observational measure used in the Mediational Intervention for Sensitizing Caregivers (MISC) and quantifies emotional (attachment-based) and cognitive (learning-based) behaviors during caregiver-child interaction. The emotional components scale ranges from 0 to 40. A higher score indicates more emotional components. Cognitive components (Focusing, Affecting, Expanding, Regulating, Rewarding) are evaluated based on their frequency along the interaction. A higher score means more frequency of those components (better outcome).
Strengths and Difficulties Questionnaire (SDQ) | Through study completion, an average of 17 months
  This is a 25 items-based scale, scored using a 3-points scale (0=not true; 2=certainly true) which provides a screening of 5 dimensions: children emotional problems, conduct problems, hyperactivity, peer-problems and pro-social behavior. All scales range from 0 to 10. A higher score means more problems (first 4 scales: worse outcome) or more pro-social behavior (last subscale: better outcome).
Achenbach System for Empirically Assessment (ASEBA) | Through study completion, an average of 17 months
  This is a very well-known 110 items-based instrument scored from 0=Not true to 2=Very often true which provides a screening in 8 clinical dimensions and 3 second order scales. Each scale has a different range. Higher scores mean higher severity of mental health problems (worse outcome).
Stirling Children's Wellbeing Scale (SCWBS) | Through study completion, an average of 17 months
  This is a 15-item scale commonly used to measure children's happiness in the last 2 weeks. Items are scored from 1 (Never) to 5 (all the time). The score ranges from 15 to 75. A higher score means more happiness (better outcome).
Child Well-Being Level (CWBL) | Through study completion, an average of 17 months
  This is a Lickert's 7-point scale to assess the child's level of happiness compared with other children of the same age. It ranges from '1=very less happy' to '8=very happier'. A higher score means more happiness (better outcome).

SECONDARY OUTCOMES:
Self-Other Mentalization Scale (SOMS) | Through study completion, an average of 17 months
  This is a 10 items-based scale answered from 1 (very less than others) to 5 (much more than others). Self- and Other- subscales scores range from 5 to 25. Higher scores mean higher mentalization capacity (better outcome)
Reflective Functioning Scale - Youth (5 items version) (RFQ-Y5) | Through study completion, an average of 17 months
  This is a shorter version of Fonagy's Reflective Function Questionnaire. It includes 5 items scored from 1 (very disagree) to 5 (very agree) and ranges from 5 to 25, being a higher score indicative of higher mentalization capacity (better outcome).
Trait Meta-Mood Scale - Children version (TMMS-C) | Through study completion, an average of 17 months
  This instrument is here used as a measure of self-mentalizing. Only the 5 item-scale of 'clarity of emotions' will be used. Items score from 1=Not at all true, to 5=Completely true. Total score ranges from 5 to 25, being a higher score indicative of higher emotional clarity (better outcome).
Big Five Questionnaire for Children and Adolescents (BFQ-NA) | Through study completion, an average of 17 months
  This questionnaire assesses the big five personality factors in young children using 65 items scored from 1=Almost always to 5=Almost never. In this study, the scale of kindness is used to score pro-social behavior, and the scale of emotional instability to score emotional dysregulation. A higher score indicates higher emotional instability (worse outcome) or higher pro-sociality (better outcome, after inverting the score).
BarOn Inventory of Emotional Intelligence for children aged 7 to 18 years old (BarOn) | Through study completion, an average of 17 months
  BarOn's scales of intra-personal (6 items) and inter-personal (12 items) scales, which are scored in 4-points scales ranging from '1=Never' to '4=Always'. The indicated subscales ranges are 4-24 and 12-48, respectively. A higher score indicates higher intelligence (better outcome).
Rosenberg's Self-Esteem Scale - Child version (RSES-C) | Through study completion, an average of 17 months
  This is a gold standard measure of self-esteem using 10 items which scored from "1=totally agree" to "4=totally disagree". After inverting the total score, which ranges from 10 to 40, a higher score means higher self-esteem (better outcome).
Battery of Socialization (BAS) | Through study completion, an average of 17 months
  The scales of social sensitivity, respect and self-control, and aggressivity, all scored using items ranging from Never (1) to Always (4), are here used to measure children's pro-social behavior. Higher scores mean higher pro-social dimensions (better outcome).
Goldberg Health Questionnaire (28 items) (GHQ-28) | Through study completion, an average of 17 months
  This is a gold standard screening of adult psychopathology in 4 areas (anxiety, depression, somatic complaints, and social dysfunction). Each area is evaluated with 7 scores from 1 to 4. Subscales range from 7 to 28. A higher score indicates a higher level of problems (worse outcome).
Difficulties in Emotional Regulation Scale (DERS) | Through study completion, an average of 17 months
  This is a gold standard to assess problems of Emotional Regulation (a key factor for mental health) using 36 items with 5 response options ranging from "1=almost never" to "5=almost always". Total score ranges 36-180. A higher score means higher emotional regulation difficulty (worse outcome).
Trait Meta-Mood Scale (24 items) TMMS-24 | Through study completion, an average of 17 months
  This instrument consists of 3 x 8-tiem subscales ('attention to emotions', 'emotional clarity' and 'emotional repair') scored with a 5-point scale ranging from "1=totally disagree" to "5=totally agree". Each scale ranges 8-40. A higher score means higher meta-mood knowledge (better outcome).
Rosenberg's Self-Esteem Scale (RSES) | Through study completion, an average of 17 months
  This is a gold standard to self-report adult self-esteem with 10 items scored from "1=totally agree" to "4=totally disagree". Total score ranges from 10 to 40. Once inverted, a higher score indicates higher self-esteem (better outcome).
Oxford Happiness Questionnaire (OHQ) | Through study completion, an average of 17 months
  This is a gold standard to assess emotional well-being based on 8 items scored from "1=totally disagree" to "6=totally agree". The scale ranges from 8 to 48. A higher score indicates higher well-being (better outcome).
Parental Reflective Function Questionnaire (PRFQ) | Through study completion, an average of 17 months
  This scale assesses parent capacity to mentalize the child (to keep the child's mind in mind) using 18 items scored from 1 (Completely disagree) to 7 (Completely agree). Total score ranges from18 to 126. A higher score indicates higher reflective parenting (better outcome).
Parental Sense of Competence Scale (PSOC) | Through study completion, an average of 17 months
  This scale consists of 10 items scored from 1 (totally disagree) to 6 (totally agree) to assess parental perceive self-competence. It ranges from 10 to 60. A higher score indicates a higher sense of self-competence in parenting (better outcome).
Parental Stress Questionnaire (PSI) | Through study completion, an average of 17 months
  This instrument consists of 36 items scored from 1 (very agree) to 5 (very disagree). Total score ranges from 36 to 180. A higher score indicates more parental stress (worse outcome).
Basic Empathy Scale (BES) | Through study completion, an average of 17 months
  This is a gold standard to assess empathy and consists of 20 items scored from 1 (totally disagree) to 5 (totally agree). Total score ranges from 20 to 100. A higher score is indicative of higher empathy (better outcome).
Maslach Burnout Inventory (MBI) | Through study completion, an average of 17 months
  This is a gold standard to assess stress at work and burnout, based on 22 items scored from 0 (Never) to 6 (Every day). Total score ranges from 22 to 132. A higher score is indicative of more stress at work or burn out (worse outcome).
Teachers' Reflective Function Questionnaire (TRFQ) | Through study completion, an average of 17 months
  This is an adaptation of the Parental Reflecting Function Questionnaire which allows to assess the mentalization stance of teachers toward their students by using 19 items scored from 1 (Completely disagree) to 7 (Completely agree). Total score ranges from 19 to 133. A higher score indicates more teachers' mentalization stance (better outcome).

OTHER OUTCOMES:
Vermunt's Learning Regulation Scale (VLRS-28) | Through study completion, an average of 17 months
  This instrument measures learning patterns, which are considered to moderate the impact of the intervention. It consists of 28 items assessing the 4 learning patterns of Vemunt's model with 4 x 7-item scales scored from 1 (Never) to 5 (Always). All 4 subscales range from 7 to 28. A higher score means a higher presence (or tendency to use) that pattern (potential moderator).
Relationship Questionnaire (RQ) | Through study completion, an average of 17 months
  This is a very brief screening scale including 4 x 7-point Lickert's to assess the 4 Bartholomew and Horowitz's relationship styles (secure, anxious-avoidant, anxious-preoccupied and disorganized) and 1 last categorical item to select the style that better identifies the participant. Attachment style could moderate the impact of parental intervention on a child's mental health. Each attachment style is scored from 1 to 7. A higher score indicates higher presence of that relationship style (potential moderator).

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Ballespí, PI, Principal Investigator — Universitat Autònoma de Barcelona
Locations (1):
- Sergi Ballespí, Barcelona, Spain/Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
The base of data will be shared through Universitat Autònoma de Barcelona (UAB) public repository